CLINICAL TRIAL: NCT01115725
Title: Phase IV Study to Evaluate the Ease of Use, Local Tolerance Safety and Effectiveness of Gonal-f® (Filled-by-Mass in a Prefilled Pen)
Brief Title: A Study to Evaluate the Ease of Use, Local Tolerance, Safety and Effectiveness of Gonal-f® (Filled-by-mass in a Prefilled Pen)
Status: Completed | Type: Observational
Sponsor: Merck KGaA, Darmstadt, Germany (Industry)
Responsible Party: Sponsor
Other Study IDs: IMP25404
Record Dates: First submitted 2010-04-30; First posted 2010-05-04 (Estimated); Last update posted 2014-07-17 (Estimated); Status verified 2012-12

CONDITIONS: Infertility
Keywords: Follitropin alfa; Fertilization in vitro; Intracytoplasmic sperm injection; Reproductive techniques, assisted
MeSH Terms: conditions — Infertility; Helping Behavior | interventions — follitropin alfa; Glycoprotein Hormones, alpha Subunit

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (1):
- Gonal-f® prefilled pen
  Interventions: Drug: Gonal-f® (follitropin alfa)

INTERVENTIONS:
Drug: Gonal-f® (follitropin alfa) — Gonal-f® (follitropin alfa) will be given once daily subcutaneously at a starting dose of 150-375 international unit per day (IU/day) by self-administered injection via a pen device for first 5 days. After Day 5, Gonal-f® dose will be adjusted according to the investigator's discretion until ovarian response observed.
  Other Names: Recombinant human follicle stimulating hormone (r-hFSH)

SUMMARY:
This is a prospective, open-label, non-comparative, multicentric Phase 4 study to evaluate the ease of use, local tolerance, safety and effectiveness of Gonal-f® (filled-by-mass in a prefilled pen) in subjects undergoing ovarian hyperstimulation for in vitro fertilization (IVF) or intracytoplasmic sperm injection (ICSI) with recombinant follicle stimulating hormone (r-FSH).

Clarification for change of study type:

The study was erroneously registered as an interventional trial on ClinicalTrials.gov between 2010 and 2012. It was shown recently that the study protocol and conduct of the study did not include any clinical interventions beyond those which are Standard Clinical Practice and the approved label for Gonal-f®. Furthermore, all other relevant study essential documentations (e.g. Informed Consent, CRF, etc.) are in line with an observational study design. As per EU regulations (Article 2(c) of Directive 2001/20/EC), this study is a 'non-interventional trial'.

DETAILED DESCRIPTION:
Treatment of subfertility and infertility by assisted reproduction technologies (ART) such as IVF and embryo transfer (ET) requires multiple follicular development to increase the number of female gametes, and the chances of a successful treatment outcome. Ovarian stimulation in IVF or ICSI currently includes suppression of endogenous luteinizing hormone (LH) secretion by administration of a gonadotropin releasing hormone (GnRH) agonist, followed by stimulation of multiple follicular development by exogenous FSH administration. When adequate follicular development is achieved, a single dose of u-hCG (urinary-human chorionic gonadotropin) is administered to mimic the endogenous LH surge and induce final oocyte maturation. Recombinant-human FSH (r-hFSH) has been shown to be superior to u-hFSH (urinary-derived FSH) in terms of requiring fewer ampoules and more efficacious in terms of number of oocytes recovered and in terms of pregnancy rates.

Recently, a new formulation of follitropin alfa has been developed as the next step in innovation in Serono capitalized on the fact that Serono recognized that follitropin alfa manufacturing was highly controlled and with a controlled specific activity that allowed filling the product by mass guaranteeing the dose being delivered. Until now follitropin alfa has been produced as a lyophilisate for injection (either as single dose or multidose applications) in glass ampoules or in glass vials and administered using syringes. Today, Gonal-f® fill-by-mass is available as a new liquid formulation that can be administered with the pen device which is prefilled and hence the subject does not have to assemble the device making it simpler to use.

OBJECTIVES

Primary objective:

To evaluate the ease-of-use of Gonal-f® (filled by mass in a prefilled pen) in subjects undergoing IVF/ICSI.

Secondary objectives:

To evaluate the local tolerance, safety and effectiveness of Gonal-f® prefilled pens.

ELIGIBILITY:
Inclusion Criteria:

* Pre-menopausal female subjects, between their 18th and 39th birthday
* Subjects with body mass index between 18-32 kilogram per square meter (kg/m^2)
* Subjects with FSH (on second day of menstrual cycle) less than 10 milli international unit per milliliter (mIU/ml)
* Subjects who required treatment with recombinant FSH for controlled ovarian hyperstimulation for IVF and/or ICSI
* Subjects who are able to communicate well with the investigator and to comply with the requirements of the entire study
* Subjects who have given written informed consent, prior to treatment, with the understanding that consent may be withdrawn by the subject at any time without prejudice

Exclusion Criteria:

* Subjects who are not pregnant or lactating
* Subjects with known allergic reaction against one of the ingredients
* Subjects with enlarged ovaries or cysts unrelated to polycystic ovaries (PCO)
* Subjects with gynecological bleeding of unknown origin
* Subjects who have ovarian, uterine, or mammary cancer
* Subjects with hyperprolactinemia
* Subjects with tumors of the hypothalamus or the pituitary gland

Ages: 18 Years to 39 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: Primary care clinic
Sampling Method: Non-Probability Sample
Enrollment: 76 (Actual)
Dates: Start 2005-11; Primary Completion 2008-06 (Actual); Study Completion 2008-07 (Actual)

PRIMARY OUTCOMES:
Convenience assessment | Post-treatment assessment (35-42 days post embryo transfer)
  Subjects' to complete ease questionnaire survey for use of Gonal-f prefilled pens.

SECONDARY OUTCOMES:
Efficacy assessments | Pre-study (within 3 months prior to study start) to days 35-42 post-hCG
  Secondary efficacy assessments include evaluation of the duration of stimulation; total amount of gonadotropins needed; number of follicles on the day of the last ultra-sound scan; estradiol (E2) on the day of the last ultra-sound scan; number of oocytes retrieved; number of oocytes fertilised; number of embryos transferred; clinical pregnancy by ultra-sound scan
Safety and tolerance assessments | First stimulation day (S1) to days 15-20 post-hCG
  Safety will be measured by the incidence and severity of adverse events (AEs) including local reactions; and incidence of ovarian hyperstimulation syndrome (OHSS)

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — Merck A.E. Hellas, an affiliate of Merck KGaA, Darmstadt, Germany
Locations (1):
- EMBRYOGENESIS IVF Unit, Athens, Kifisias aV, Greece